CLINICAL TRIAL: NCT02859571
Title: Continuous Versus Intermittent Oxytocin for Induction of Labor: A Randomized Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, medical doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 152
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Intemittant, Continue, Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous oxytocin (Active Comparator): oxytocin will be used at a starting dose of 1-2 mIU/min and the dose will be increased by 2 mIU/min at every 15 minutes until regular contractions will be obtained at a rate of 3-5 contractions in a 10-minute period. The maximum dose of oxytocin will 40 mIU/min and oxytocin will be administered until delivery.
  Interventions: Drug: Oxytocin
- intermittent oxytocin (Experimental): oxytocin will be discontinued when cervical dilation will 5 cm and 2 hours after discontinuation oxytocin will be reused at a starting dose of 1-2 mIU/min and will be increased as the same protocol will be used for continuation oxytocin group.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
This study evaluates continuous oxytocin versus intermittent oxytocin for induction of labor at term. Half of participants will be taken continuous oxytocin, while the other half will be taken intermittent oxytocin.

DETAILED DESCRIPTION:
In the continuous oxytocin group, traditional treatment of oxytocin used at a starting dose of 1-2 mIU/min and the dose was increased by 2 mIU/min at every 15 minutes until regular contractions obtained at a rate of 3-5 contractions in a 10-minute period. The maximum dose of oxytocin was 40 mIU/min and oxytocin was administered until delivery. In the intermittent group, oxytocin was discontinued when cervical dilation was 5 cm and 2 hours after discontinuation oxytocin was reused at a starting dose of 1-2 mIU/min and was increased as the same protocol used for continuation oxytocin group.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy,
* 37≤ weeks of gestational age ,
* vertex presentation,
* women with cervical dilation 3 cm
* no contraindication to vaginal delivery.

Exclusion Criteria:

* fetal malpresentation,
* multifetal pregnancy,
* more than three contractions in 10 minutes,
* contraindications to oxytocin,
* a category II or III fetal heart rate pattern,
* fetal anomaly,
* fetal demise
* women with immediate delivery indications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
induction-to-delivery time | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: evrim bostanci ergen, Principal Investigator — Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Locations (1):
- Zeynep Kamil Maternity and Children's Training and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bor P, Ledertoug S, Boie S, Knoblauch NO, Stornes I. Continuation versus discontinuation of oxytocin infusion during the active phase of labour: a randomised controlled trial. BJOG. 2016 Jan;123(1):129-35. doi: 10.1111/1471-0528.13589. Epub 2015 Aug 26. PMID 26309128
- [Background] Ozturk FH, Yilmaz SS, Yalvac S, Kandemir O. Effect of oxytocin discontinuation during the active phase of labor. J Matern Fetal Neonatal Med. 2015 Jan;28(2):196-8. doi: 10.3109/14767058.2014.906573. Epub 2014 Apr 9. PMID 24646336